CLINICAL TRIAL: NCT02880150
Title: Physiological Characteristics of High Altitude Climbers
Acronym: ALTIPERF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013-A00629-36; ALTIPERF (Other: Grenoble University Hospital)
Record Dates: First submitted 2013-10-21; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Hypoxia; Exercise; Sport Performance
Keywords: elite climbers; near infrared spectroscopy
MeSH Terms: conditions — Hypoxia; Motor Activity | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elite climbers (Other): Elite climbers selected in a national group for their previous performances at high altitude
  Interventions: Other: Stress test
- Sea level sportsmen (Other): Control group with similar anthropometric, age, gender and maximal normoxic oxygen consumption that the elite climber group
  Interventions: Other: Stress test

INTERVENTIONS:
Other: Stress test

SUMMARY:
Climbing at high altitude and tolerating hypoxic environment require specific physiological adaptations. Large intersubjects differences exist regarding the ability to adapt to high altitude and hypoxia. The present study aims to characterise the physiological responses to hypoxia in a group of elite climbers by comparison to sea level athletes. We hypothesised that elite climbers would show better physiological responses to hypoxia and more preserved performances compared to sea level.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40
* Member of the national high altitude climbing group

Exclusion Criteria:

* Any diseases incompatible with hypoxic exposure, exercise testing
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Performance reduction in hypoxia versus normoxia | Day one on the evaluation day
  Difference in maximal cycling power output between the normoxic and the hypoxic exercise test

SECONDARY OUTCOMES:
Near infrared signals during exercise | Day one on the evaluation day
  Differences in cerebral and muscle TOI during exercise between the normoxia and the hypoxic exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble University Hospital, Grenoble, France

REFERENCES:
- [Background] Verges S, Rupp T, Jubeau M, Wuyam B, Esteve F, Levy P, Perrey S, Millet GY. Cerebral perturbations during exercise in hypoxia. Am J Physiol Regul Integr Comp Physiol. 2012 Apr 15;302(8):R903-16. doi: 10.1152/ajpregu.00555.2011. Epub 2012 Feb 8. PMID 22319046